CLINICAL TRIAL: NCT05847777
Title: Correlation Between Maxillary Sinus (Linear and Volumetric Measurements) and Midface Width Using CBCT A Cross Sectional Study
Brief Title: Correlation Between Maxillary Sinus (Linear and Volumetric Measurements) and Midface Width Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Hassan, Assistant lecturer PhD Candidate, Cairo University
Other Study IDs: ORAD3 -3 -1
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Cone-beam Computed Tomography; Maxillary Sinus; Midface; Volumetric Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: CBCT — cone beam computer tomography

SUMMARY:
The objective of this study will be To assess the correlation of the 2-D and volumetric maxillary sinus dimensions with the linear measurement of the mid-face width in adult Egyptian individuals. The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes. The following radiographic examination will be done in Oral and Maxillofacial Radiology Department, Faculty Dentistry, Cairo University. semiautomated segmentation will be performed for the maxillary sinus in both side and then linear and volumetric measurements will be assessed for each sinus. Also the width of midface will be assessed.

DETAILED DESCRIPTION:
The objective of this study will be To assess the correlation of the 2-D and volumetric maxillary sinus dimensions with the linear measurement of the mid-face width in adult Egyptian individuals. The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes. The following radiographic examination will be done in Oral and Maxillofacial Radiology Department, Faculty Dentistry, Cairo University. semiautomated segmentation will be performed for the maxillary sinus in both side and then linear and volumetric measurements will be assessed for each sinus. Also the width of midface will be assessed.

CBCT images will be analysed using Mimics software (version 21.0; Materialise, Leuven, Belgium). To measure volumes of the maxillary sinuses, thresholding will be applied with minimum and maximum limits of - 1024 HU and - 526 HU, respectively. The maxillary sinus will be cropped using the software's "edit masks" tool along the following borders: around the bone structure and narrowest space of the ostium between the infundibulum and the uncinate process After this, three-dimensional (3D) models of the sinuses will be created and the volumes of the right and left sinuses will be calculated separately by giving different colors to the sinuses of the same patient.

Slice thickness will be maintained at 0.4 mm as a standard for further 2-D and 3-D reconstruction.

All maxillary sinus measurements will be performed separately on the left and right sides.

For the maxillary sinus linear 2D measurements, each scan will be assessed for:

Maximal vertical diameter (maximal height) of the maxillary sinus (MSH) involves the longest distance from the lowest point of the inferior wall to the highest point of the superior wall in the adjusted sagittal image.

Maximal horizontal diameter (maximal width) of the maxillary sinus (MSW) involves the longest distance perpendicular from the most prominent point of the medial wall to the most prominent point of the lateral wall on the adjusted axial image.

Maximal anteroposterior diameter (maximal length) of the maxillary sinus (MSL) involves the longest distance from the most anterior point of the anterior wall to the most posterior point of the posterior wall on the adjusted the axial image.

To measure the midface width on CBCT adjusted coronal image, the most lateral and inferior point of the maxillozygomatic suture (zm point) on both sides will be detected and measure the distance between them.

To measure one side maxillary width, the distance between (zm point) of one side to mid palatine will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of adult Egyptian patients, males and females, with age range between 18 and 50 years old. Patients will be divided into two age groups (group 1 less than or equal 30 years old, group2 more than 30 years old).
* CBCT scans of patient without previous orthodontic treatment.
* CBCT scans without any other treatment that might interfere with the natural course of maxillomandibular growth and development.

Exclusion Criteria:

* Scans with maxillary pathologies like (tumors, odontogenic lesions, bone lesions).
* Patients with traumatic injuries or fractures affecting the maxillary sinus.
* Patients with missing upper premolar or molar teeth in one side or both sides.
* Patients with skeletal asymmetries, craniofacial traumas and developmental anomalies such as palatal cleft.
* Images of low-resolution quality.
* Distortion of images or presence of any artifacts.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: CBCT maxillofacial scans belonging to Egyptian individuals will be examined
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Maxillary sinus linear measurements with width of midface | 1 year
Correlation between Maxillary sinus volumetric measurements with width of midface | 1 year

SECONDARY OUTCOMES:
Correlation between Maxillary sinus volumetric measurement with mandibular body length | 1 year
Maxillary sinus volume dimensions with age variables | 1 year
Maxillary sinus volume dimensions with sex variables | 1 year

REFERENCES:
- See also: Related Info — https://drive.google.com/file/d/1OiBb70gpr7PXZVQej9fhbzCL7ttIQvlA/view?usp=share_link